CLINICAL TRIAL: NCT04704609
Title: Imaging Quantification of Inflammation (IQI)
Acronym: IQI
Status: Active, not recruiting | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Santen Inc. (Industry)
Responsible Party: Principal Investigator, Sunil Srivastava, Principle Investigator, The Cleveland Clinic
Other Study IDs: 17-1258
Record Dates: First submitted 2020-10-21; First posted 2021-01-11 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Imaging Analysis of patients with uveitis: Any patient with a diagnosis of uveitis, who is deemed active or recently active (6 months) by a uveitis specialist
  Interventions: Other: Standard of Care Imaging

INTERVENTIONS:
Other: Standard of Care Imaging — We are collecting imaging that is standard of care for uveitis patients

SUMMARY:
1. Perform observational study utilizing real-time quantification of ocular inflammation to determine minimal important change.

Prospective use of changes in imaging quantification of inflammation (IQI) scores in determining treatment decisions both utilizing novel FA viewer software.

DETAILED DESCRIPTION:
1. Perform observational study utilizing real-time quantification of ocular inflammation to determine minimal important change.

   In our current experiments, we have calculated reliability measurements including the standard error of measurement (SEM) for our software tools. Our hypothesis is that the minimal important change seen clinically will be at least equal to the standard error of measurement. This is based on previous work observing the use of SEM as the minimal important change on outcome scales.56-58 We hypothesize that changes in the imaging quantification of inflammation scores (IQI) of greater than SEM, will lead to observed changes in visual function.

   To test our hypothesis we will prospectively observe 25 patients with uveitis who are either active or were recently active in the previous 6 months. All of the patients will have standard clinical exams at baseline and image quantification of their inflammation using OCT, OCTA and UWFFA (if needed). At baseline, ETDRS vision, contrast sensitivity, hand held electroretinography and a visual function questionnaire (NEI-VFQ 25) will be administered. Patients will be followed for 6 months. During follow-up repeat imaging quantification of inflammation will be performed along with standard examinations, visual acuity and contrast sensitivity measurements and hand held ERG. At the final visit, all tests will be repeated. Data collected will be analyzed using statistical software package. Correlations between changes in imaging quantification of inflammation scores and changes in visual acuity, clinical grades of inflammation, visual function scores and contract sensitivity will be calculated. Expected outcomes include confirmation that a change in IQI scores greater than standard error of measurement will result in a clinically meaningful change. We now would have a definition of improvement and worsening based on changes in IQI scores.

   Image acquisition protocols will depend on subtype of uveitis. In those with anterior uveitis, only OCT, OCTA and anterior segment OCT will be obtained by study staff. In those with posterior segment uveitis, UWFFA will be obtained as part of standard of care.
2. Prospective use of changes in imaging quantification of inflammation (IQI) scores in determining treatment decisions As the above experiment will have defined the scores required for improvement and worsening, we will assess the use of these tools in making clinical treatment decisions. We hypothesize that clinician use of imaging based quantification of inflammation (IQI) scores will impact clinical decision making. We intend to test our hypothesis with the following experiment. 25 patients with active or recently active (within 6 months) uveitis will be enrolled in a prospective study. At baseline patients will have standard of care examinations performed and IQI scores will be acquired using OCT, OCTA and UWFFA. Patients will be followed over a period of 1 year. At subsequent follow-up visits, IQI scores will be obtained. Prior to the clinician examining the patient, the IQI scores will be reviewed and compared to the previous visit(s). The clinician will then fill out a survey form indicating if (s)he would treat based on IQI scores, observe based on IQI scores, or can't decide by IQI alone. At this point the clinician would then examine the patient and fill out a second questionnaire evaluating whether (a) clinical exam agreed with IQI, (b) clinical exam did not agree with IQI (c) clinical exam did not pick up changes that IQI found. The patient will then be treated by clinical judgment with clinical exam and IQI scores available to the physician. The data collected will be analyzed using a statistical software package. (SAS) Percentage agreement, correlation between exam results and IQI scores will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a diagnosis of uveitis, who is deemed active or recently active (6 months) by a uveitis specialist

Exclusion Criteria:

* Poor view in fundus in both eyes which precludes image acquisition in those with posterior uveitis
* Those with posterior uveitis, any allergy to fluorescein
* Corneal opacities which prevent image acquisition
* Inability to sign consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ocular inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-09-22 (Actual); Primary Completion 2027-04-20 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Real Time Quantification of Ocular inflammation | 6 months
  Perform observational study utilizing real-time quantification of ocular inflammation to determine minimal important change using FA viewer software.

SECONDARY OUTCOMES:
Scoring ocular inflammation for clinical use | 6 months
  Prospective use of changes in imaging quantification of inflammation (IQI) scores in determining treatment decisions

CONTACTS AND LOCATIONS:
Overall Officials: Sunil K Srivastava, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation Cole Eye Institute, Cleveland, Ohio, United States